CLINICAL TRIAL: NCT02258763
Title: Pneumonia in Children: Aetiology, Ideal Antibiotic Duration, Quality of Life
Brief Title: Trial on the Ideal Duration of Oral Antibiotics in Children With Pneumonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: Menzies School of Health Research (Other)
Responsible Party: Principal Investigator, Anna Marie Nathan, Consultant and Associate Professor, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RP026-14HTM
Record Dates: First submitted 2014-09-23; First posted 2014-10-07 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Pneumonia
Keywords: Pneumonia; Child; Outcome; Antibiotics; Etiology
MeSH Terms: conditions — Pneumonia | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amoxicillin-Potassium Clavulanate (Experimental): Patient will be on amoxicillin-clavulanate 22.5mg/kg/dose bd for 10 days
  Interventions: Drug: Amoxicillin-Potassium Clavulanate Combination
- Placebo (Active Comparator): Patient will be on amoxicillin-clavulanate 22.5mg/kg/bd for 3 days followed by another 7 days of placebo medication given at the same dose and frequency
  Interventions: Drug: Amoxicillin-Potassium Clavulanate Combination; Drug: Placebo

INTERVENTIONS:
Drug: Amoxicillin-Potassium Clavulanate Combination — Oral antibiotic for 10 days
  Other Names: Augmentin; Clomovid; Co-amoxiclav
Drug: Placebo — Placebo made to look like the study drug-main ingredient sugar syrup made by the pharmacy department in the hospital In the placebo arm, patient will be given 3 days of antibiotic followed by 7 days of placebo
  Other Names: Placebo arm
  Arms: Placebo

SUMMARY:
To determine, in children hospitalized with pneumonia, if an extended duration of oral antibiotics (10 days) will be superior to a shorter duration (3 days) of antibiotics in improving clinical outcomes.

Secondary Aims:

1. Describe the prevalence of respiratory viruses and bacteria at presentation.
2. Investigate the depression, anxiety and stress scores (DASS21) and quality of life scored (QOL) by parents of the children during admission, pre-discharge and post discharge and at follow-ups.

DETAILED DESCRIPTION:
Introduction:

Pneumonia is the single largest cause of death in children less than 5 years old and these are preventable deaths.[1,2] It is also an important cause of morbidity , especially when it is recurrent or severe as it may be linked with future adult lung disease.[3] Determining the aetiology of pneumonia is difficult in children who cannot produce satisfactory sputum for culture. Hence the reliance on molecular methods like polymerase chain reaction (PCR) and Enzyme immunoassays(EIA) looking at serological rise to determine the true aetiology of pneumonia is important especially in the era where mixed infections are common and may be associated with severe infections.

There is currently no information on the suitable duration of antibiotics for uncomplicated severe community acquired pneumonia (CAP). There is also rampant overuse of antibiotics that results in poor compliance and significant side effects.

There is little information on the QOL of the child with severe pneumonia and his parent. It is important to have a holistic approach to medicine hence the importance of analyzing the burden and social issues associated with children admitted with pneumonia.

As opposed to adults, children cannot produce sputum (lower respiratory sample) appropriate for culture which is the traditional method of identifying the causative bacteria. Identification of bacteria in nasopharyngeal secretions (upper respiratory sample) does not equate to that organism causing the infection as the upper airway of a child is often colonized by bacteria. Detecting the organism in blood identifies it as the causative organism. However, blood culture has a very low yield in children with pneumonia and polymerase chain reaction (PCR) is much more sensitive at detecting bacteria in blood and hence it will markedly improve the ability to determine infecting organism.

Development of our own in-house bacterial PCR kit which will detect several different bacteria in blood is planned in this study. We already have an in-house viral PCR kit and the ability to detect atypical bacteria via EIA. Currently there is an international study (Pneumonia Etiology Research for Child Health [PERCH]) looking at aetiology of pneumonia, but this study only involves 2 Asian countries (Thailand and Bangladesh)[5]. In Malaysia, in 2011 there was a study that looked at pneumococcal isolates and antibiotic sensitivity patterns on invasive pneumococcal disease only[6]. There are also studies that look at viral aetiology of pneumonia[7]. Hence information on aetiology of pneumonia is skewed to those involving vaccine associated organisms and use of nasopharyngeal secretions(NPS) to detect viruses..

The evidence for appropriate duration of antibiotics that should be used in hospitalized children with pneumonia is scarce. A randomized controlled trial comparing traditional duration of antibiotics (≥ 7 days) versus shorter duration of antibiotics < 7 days) is what we think is necessary. There are no studies looking at duration of antibiotics in children with severe uncomplicated pneumonia. We hypothesize that there is no need for a longer duration of antibiotics which are only associated with poor compliance and unnecessary side-effects.

Finally, there is little data on quality of life in children and parents during and after a pneumonic episode. It is important to measure the impact of such a common disease on both parent and patient as well as to assess the impact of medical management on QOL so as to have a more holistic approach to medicine. Two previous studies have looked at QOL. One was a study comparing all acute diseases to chronic diseases[8]. The other looked at CAP but without the use of structured questionnaires[9]

Methodology

Randomized, Double Blind, Placebo Controlled Trial Children aged 3 months till <5 years old Admitted to University Malaya Medical Centre (UMMC) hospital with a severe community acquired pneumonia Eligibility Ages Eligible for Study: 3 Months to 59 Months Genders Eligible for Study: Both

Inclusion Criteria:

Children admitted with severe pneumonia as defined by the presence of all the following as defined as below:

* 3 months to 59 months old
* History of cough and/or shortness of breath Unwell for <= 7 days
* Increased respiratory rate ( ≥ 50/min if ≤12 months old, ≥ 40/min)
* Any of the following signs/symptoms are present at examination that would necessitate admission: chest retractions, cyanosis, saturation< 92% on air, poor feeding or lethargy
* Documented fever (axillary /central temp ≥ 38/38.5°C) within 24 hrs of admission
* Abnormal chest radio graph(CXR) with presence of alveolar infiltrates
* Responds to IV antibiotics by the first 72 hrs and able to go home with oral antibiotics i.e. no more hypoxia and afebrile and reduced respiratory symptoms

Exclusion Criteria:

Children who (a) are transferred from another hospital (b) refuse blood taking (c) have a doctor diagnosis of asthma or recurrent wheezing illness (d) have a diagnosis of bronchiolitis i.e. wheezing in a child with a CXR with no consolidation (e) do not have an acute illness ( ie >7 days) (f) are unable to come for follow-up (g) do not have community acquired pneumonia e.g. aspiration pneumonia (h)have a complicated pneumonia with effusion, pneumothorax, clinical suspicion of necrotizing pneumonia (i)require paediatric intensive care unit (PICU) admission or use of non-invasive ventilation (j)significant comorbidities that can increase the risk of having a complicated pneumonia- (k) need other antibiotics like anti-staph or macrolides (l)have an extra-pulmonary infection e.g. meningitis (m)are allergic to penicillin (n) are unable to tolerate oral antibiotics and (o)have underlying illness that can predispose to recurrent pneumonia

Randomized, Double Blind, Placebo Controlled Trial Children aged 3 months till <5 years old Admitted to UMMC hospital with a severe community acquired pneumonia Informed signed consent will be obtained from parents first. All children will have full blood count and CXR taken

Additional blood and urine as detailed below will also be taken:

a. Blood for PCR -streptococcus pneumoniae, staphylococcus aureus, Haemophilus influenzae, Mycoplasma pnuemoniae, Chlamydia pneumoniae will be taken.

NPS for respiratory bacteria and viruses (by culture and PCT-similar as above) All these samples will be tested in our hospital laboratory. If samples cannot be processed immediately, they will be stored in a -80 deg C freezer except for the NPS for bacterial culture.

All data will be collected at enrollment and at each follow-up visit on a standardized data sheet. Baseline demographic data( age, gender, address, ethnicity, household size, income, parent education, caregivers, household appliances) and medical information( birth history, breastfeeding and weaning, growth, immunization, smoke exposure, co-morbidity, daily hospitalization information) will be obtained from parents and medical charts. CXRs and routine blood test results will also be recorded.

Quality of life, stress level, severity of illness , of parents and children with pneumonia, will be assessed at these time points too: during their admission (average of 3-5 days) and during follow-ups( average at, 4 weeks, 3 months(phone call only with no questionnaire administered), 6 months, 1 year post their pneumonic episode) using the following questionnaires-Paediatric proxy cough quality of life-8 (PCQOL-8), Canadian Acute Respiratory Illness and Flu Scale (CARIFS) (in hospital only), cough diary( at home, daily for 1 month),Depression Anxiety Stress Scale 21( DASS21).

The PCQOL-8 and DASS21 have been translated and validated in Bahasa Melayu. The CARIFS and the cough diary was recently translated in Bahasa Melayu and piloted for the purpose of this study.

Treatments will be administered only after at least 48-72 hrs of intravenous(IV) antibiotics ( penicillin/ampicillin/ amoxicillin-clavulanate acid/cefuroxime) and the patients are ready for discharge : afebrile, improved respiratory symptoms and signs, saturation > 92% in air and ready to be converted to oral antibiotics.

Arm 1: Twice a day oral amoxicillin-clavulanate (22.5mg/kg/dose) for 10 days Arm 2: Twice a day oral amoxicillin-clavulanate (22.5mg/kg/dose) for 3 days followed by oral placebo for 7 days The random treatments will be allocated via computer generated number sequence and will be supervised by a statistician.

All medications will be prepared and dispensed by the pharmacy department in suspension form. The appearance of the placebo will be similar to the active medication. Investigators and subjects will be blinded.

At discharge, parents will be asked to fill up a daily cough diary at home. Treatment failure/exit criteria will be fulfilled if any of the following occur: death, recrudescence of fever ≥38 °C (axilla) with respiratory signs of pneumonia, hypoxaemia < 92% on air), need for antibiotic treatment, new CXR changes.

On discharge, children will be followed up at regular intervals of 4 weeks, 3 moths(phone call), 6 months and 1 year, to ensure they are well and also to detect residual or recurring respiratory symptoms i.e. presence of cough/breathlessness/fever, recrudescence of pneumonia and other respiratory illness, fever and upper respiratory tract infection(URTI), growth, need for unscheduled healthcare visits for respiratory symptoms, need for antibiotic treatments for respiratory/upper airway symptoms, abnormal physical findings, over a period of 1 year post-discharge from hospital. Adverse effects of antibiotics e.g. vomiting, diarrhoea, rash and adherence (returned empty bottles) to medication will be recorded.

CXR will be repeated at 4 weeks and at 1 year(if clinically indicated). These will be scored by a radiologist who will be masked to allotted treatment.

At 12 months, if the age allows it, children will be asked to perform lung function tests.

During these follow-ups they will be given questionnaires: PCQOL-8, DASS21. At the 4 week discharge, CXR as well as blood and NPS will be collected for testing for bacterial and viral organisms. At 4 weeks, daily cough diaries will be collected back and reviewed.

Sample size calculation is based on the primary aim. We expect a 20% superiority difference in the extended antibiotic regime and assuming a 20% drop-out, sample size should be 204 children (102 in each arm).

Data will be presented in accordance with the CONSORT guidelines on reporting on RCTs. Analysis will be done by Dr. Rafdzah, a statistician. An intention to treat approach will be used for all analyses. For the primary aim i.e. the clinical outcome of the different antibiotic durations, the main outcomes being looked at are (a) clinical cure-complete resolution of symptoms and signs at 4 weeks ,(b) proportion of children without chronic respiratory symptoms or signs at the 12 month follow-up , using odds ratio(95%CI) with logistic regression and linear regression. For continuous variables, t-tests and Mann-Whitney tests will be used depending on the normality of the data. A Kaplan-Meier curve will be constructed for each group for the time to next respiratory illness and hospitalization and proportions will be compared by regression models. For prevalence of respiratory pathogens, point prevalence will be reported on and multivariable logistic regression adjusting for baseline carriage and antibiotic resistance will examine the effects of treatment duration on the different organisms particularly Streptococcus pneumoniae and Haemophilus influenzae and Staph aureus.

ELIGIBILITY:
Inclusion Criteria:

Children admitted with severe pneumonia as defined by the presence of all the following as defined as below:

* 3 months to 59 months old
* History of cough and/or shortness of breath
* Unwell for <= 7 days -Increased respiratory rate ( ≥ 50/min if ≤12 months old, ≥ 40/min) or retractions,-
* Any of the following signs/symptoms are present at examination that would necessitate admission: chest retractions, cyanosis, saturation< 92% on air, poor feeding or lethargy
* Documented fever (axillary /central temp ≥ 38/38.5°C) within 24 hrs of admission
* Abnormal CXR with presence of alveolar infiltrates
* Responds to IV antibiotics by the first 72 hrs and able to go home with oral antibiotics i.e. no more hypoxia and afebrile and reduced respiratory symptoms

Exclusion Criteria:

Children who (a) are transferred from another hospital (b) refuse blood taking (c) have a doctor diagnosis of asthma or recurrent wheezing illness (d) have a diagnosis of bronchiolitis i.e. wheezing in a child with a CXR with no consolidation (e) not acute illness ( ie >7 days) (f) unable to come for follow-up (g) not community acquired pneumonia e.g. aspiration pneumonia (h)complicated pneumonia with effusion, pneumothorax, clinical suspicion of necrotizing pneumonia (i)PICU admission or use of Non-invasive ventilation (j)significant comorbidities that can increase the risk of having a complicated pneumonia- (k) need for use of other antibiotics like anti-staph or macrolides (l)extra-pulmonary infection e.g. meningitis (m)allergy to penicillin (n) unable to tolerate oral antibiotics (o) underlying illness that can predispose to recurrent pneumonia

-

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2014-11; Primary Completion 2017-11 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Clinical cure | 30 days
  Complete resolution of symptoms. No treatment failure or exit failure i.e. need for antibiotics or readmission into hospital for a respiratory condition

SECONDARY OUTCOMES:
Quality of life of child and parent | on admission, at discharge, at follow-ups( 4 weeks, 6 months and 1 year)
  Severity of cough by using the translated and validated PCQOL-8 to assess impact of cough on the child and parent.
Impact of pneumonia on the parent | on admission, at discharge, at follow-ups(average 1 week, 4 weeks, 6 months and 1 year)
  Using the translated and validated DASS21 on parents
Severity of pneumonia | during the admission which expected duration will be 5 days, daily twice a day to do the questionnaires
  Using the translated and validated the Canadian Acute Respiratory Influenza Scale(CARIFS)
Adverse effects | at 4 weeks follow-up
  Treatment related adverse effects of antibiotics e.g. diarrhoea, vomiting
Time to next hospitalisation or visit to healthcare unit | during the one year post pneumonic episode; patient will be seen on an avearge of 1 week, 4 weeks, 6 months and 1 year
  Time to the next hospitalization or visit to the doctor for respiratory symptoms
Number hospitalised for pneumonia or unscheduled healthcare visits | during the one year post pneumonic episode; patient will be seen on an avearge of 1 week, 4 weeks, 6 months and 1 year
  proportion of children hospitalised for respiratory illness or need for unscheduled healthcare visits
Bacterial isolates | at the 4 weeks appointment
  Bacterial isolates: resistance pattern, resolution or persistence. Viral isolates: positive or negative These will be assessed at admission and 4 weeks post-discharge
Radiological resolution | at the 4 weeks appointment
  Radiological resolution and correlation with respiratory symptoms
Prevalence of chronic respiratory symptoms and signs post pneumonia | during the one year post pneumonic episode; patient will be seen on an avearge of 1 week, 4 weeks, 6 months and 1 yea
  Presence of respiratory symptoms and signs e.g. cough, failure to thrive, reduced effort tolerance, clubbing, persistent respiratory signs
Severity of cough during 4 weeks post-discharge | at the 4 weeks appointment, cough diary which will be done by parents daily from discharge
  Using the visual scale cough diary

OTHER OUTCOMES:
Cost effective analysis of long vs short course of antibiotics for pneumonia | at the 4 weeks appointment
  To see if the extended antibiotic course is cost effective

CONTACTS AND LOCATIONS:
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Lembah Pantai, Malaysia

REFERENCES:
- [Result] Rudan I, Boschi-Pinto C, Biloglav Z, Mulholland K, Campbell H. Epidemiology and etiology of childhood pneumonia. Bull World Health Organ. 2008 May;86(5):408-16. doi: 10.2471/blt.07.048769. PMID 18545744
- [Result] Walker CLF, Rudan I, Liu L, Nair H, Theodoratou E, Bhutta ZA, O'Brien KL, Campbell H, Black RE. Global burden of childhood pneumonia and diarrhoea. Lancet. 2013 Apr 20;381(9875):1405-1416. doi: 10.1016/S0140-6736(13)60222-6. Epub 2013 Apr 12. PMID 23582727
- [Result] Chang AB, Byrnes CA, Everard ML. Diagnosing and preventing chronic suppurative lung disease (CSLD) and bronchiectasis. Paediatr Respir Rev. 2011 Jun;12(2):97-103. doi: 10.1016/j.prrv.2010.10.008. Epub 2010 Dec 4. PMID 21458737
- [Result] Trenholme AA, Byrnes CA, McBride C, Lennon DR, Chan-Mow F, Vogel AM, Stewart JM, Percival T. Respiratory health outcomes 1 year after admission with severe lower respiratory tract infection. Pediatr Pulmonol. 2013 Aug;48(8):772-9. doi: 10.1002/ppul.22661. Epub 2012 Sep 19. PMID 22997178
- [Result] Gilani Z, Kwong YD, Levine OS, Deloria-Knoll M, Scott JA, O'Brien KL, Feikin DR. A literature review and survey of childhood pneumonia etiology studies: 2000-2010. Clin Infect Dis. 2012 Apr;54 Suppl 2(Suppl 2):S102-8. doi: 10.1093/cid/cir1053. PMID 22403223
- [Result] Yasin RM, Zin NM, Hussin A, Nawi SH, Hanapiah SM, Wahab ZA, Raj G, Shafie N, Peng NP, Chu KK, Aziz MN, Maning N, Mohamad JS, Benjamin A, Salleh MA, Zahari SS, Francis A, Ahmad N, Karunakaran R. Current trend of pneumococcal serotypes distribution and antibiotic susceptibility pattern in Malaysian hospitals. Vaccine. 2011 Aug 5;29(34):5688-93. doi: 10.1016/j.vaccine.2011.06.004. Epub 2011 Jun 30. PMID 21723357
- [Result] Chan PW, Goh AY, Chua KB, Kharullah NS, Hooi PS. Viral aetiology of lower respiratory tract infection in young Malaysian children. J Paediatr Child Health. 1999 Jun;35(3):287-90. doi: 10.1046/j.1440-1754.1999.00359.x. PMID 10404452
- [Result] Kulpeng W, Sornsrivichai V, Chongsuvivatwong V, Rattanavipapong W, Leelahavarong P, Cairns J, Lubell Y, Teerawattananon Y. Variation of health-related quality of life assessed by caregivers and patients affected by severe childhood infections. BMC Pediatr. 2013 Aug 13;13:122. doi: 10.1186/1471-2431-13-122. PMID 23941314
- [Result] Shoham Y, Dagan R, Givon-Lavi N, Liss Z, Shagan T, Zamir O, Greenberg D. Community-acquired pneumonia in children: quantifying the burden on patients and their families including decrease in quality of life. Pediatrics. 2005 May;115(5):1213-9. doi: 10.1542/peds.2004-1285. PMID 15867027
- [Result] Edmond K, Scott S, Korczak V, Ward C, Sanderson C, Theodoratou E, Clark A, Griffiths U, Rudan I, Campbell H. Long term sequelae from childhood pneumonia; systematic review and meta-analysis. PLoS One. 2012;7(2):e31239. doi: 10.1371/journal.pone.0031239. Epub 2012 Feb 22. PMID 22384005
- [Result] Jimenez Ortega AI, Lopez-Neyra A, Sanz Santiago V, Alvarez-Coca J, Villa Asensi JR. [Pulmonary function in children following community-acquired pneumonia contracted at pre-school age]. An Pediatr (Barc). 2011 Nov;75(5):314-9. doi: 10.1016/j.anpedi.2011.05.002. Epub 2011 Jul 31. Spanish. PMID 21684825